CLINICAL TRIAL: NCT05658965
Title: Intérêt de l'électroencéphalogramme précoce en Chirurgie de Cardiopathie congénitale Pour prédire la Survenue de Troubles du neurodéveloppement
Brief Title: KIDSHEART AND BRAIN : Early EEG Surgery Congenital Heart Disease Predict Onset of Neurodevelopmental Disorders
Acronym: KHB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2021_0160; 2022-A00335-38 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2022-12-12; First posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-11

CONDITIONS: Neurodevelopmental Disorders; Congenital Cardiomyopathy
Keywords: EEG; Neurodevelopmental Disorders; Congenital Cardiomyopathy; Orality Disorders
MeSH Terms: conditions — Neurodevelopmental Disorders; Cardiomyopathy, infantile histiocytoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Congenital cardiopathy are frequent malformations (1/100 birth). The progress of surgery permit a survival rate at the adult age of more than 90%. The long terms consequences must be taken in account and the nerodevelopmental disorders are in first place (intelectual deficiency, autism spectrum disorders, or attention disorders) and presents in 30 to 60% of the patients (Calmant, 2015). The impact can be important on the scolarity, the studies, the professional activity and finaly on the quality of life of the patients becomming adults.

The identification of the risk factors on surgery period should permit to propose the most adapted follow-up to the specifics needs of each patients.

On the scientific plans, the identification of early markers on brain dammage on EEG should permit to better apprehend the physiopathologic mecanisms involved.

DETAILED DESCRIPTION:
Interest of early EEG on congenital cardiopathy surgery to predict the neurodevelopmental disorders occurence.

Congenital cardiopathy are frequent malformations (1/100 birth). The progress of surgery permit a survival rate at the adult age of more than 90%. The long terms consequences must be taken in account and the nerodevelopmental disorders are in first place (intelectual deficiency, autism spectrum disorders, or attention disorders) and presents in 30 to 60% of the patients (Calmant, 2015). The impact can be important on the scolarity, the studies, the professional activity and finaly on the quality of life of the patients becomming adults.

The identification of the risk factors on surgery period should permit to propose the most adapted follow-up to the specifics needs of each patients.

On the scientific plans, the identification of early markers on brain dammage on EEG should permit to better apprehend the physiopathologic mecanisms involved.

ELIGIBILITY:
Inclusion Criteria:

* Child of less than 1 year admitted for cardiac surgery on extracorporal circulation on the CHU of Lille during the study period.
* Child with congenital cardiopathy with necessity to be operated before 1 year old.

Exclusion Criteria:

* Child with no necessity of surgery before 1 year old.
* Medical history of cardiac surgery.
* Refusal of consent by the parents.
* No social security.
* Child not operated on the CHU of LILLE.

Ages: 1 Day to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children of less than 1 year suffering of congenital cardiopathy admitted for cardiac surgery on extracorporal circulation on the CHU of Lille.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2025-10-10 (Estimated); Study Completion 2025-10-10 (Estimated)

PRIMARY OUTCOMES:
Interest of pre and post surgery EEG on neurodevelopmental disorders | Age of patient : 24 Months
  Evaluation of the interest of pre and post surgery EEG in the prediction of neurodevelopmental disorders on patients operated of congenital cardiopathy before the age of 1 year old.

SECONDARY OUTCOMES:
Association between orality disorders and neurodevelopmental disorders | Age of patient : 24 Months
  Association between the presence of pre surgery and 1 year old orality disorder and occurence of neurodevelopmental disorders.
Interest of post surgery EEG neurodevelopmental disorders at 24 months old | Age of patient : 24 Months
  Evaluation of the interest of 24 months old post surgery EEG in the prediction of neurodevelopmental disorders on patients operated of congenital cardiopathy before the age of 1 year old, having a normal pre surgery EEG.

CONTACTS AND LOCATIONS:
Overall Officials: Flavien GAUTRON, CRA, Study Chair — CHU de Lille; Gaëlle GUYOT, CRA, Study Chair — CHU de Lille
Locations (1):
- CHU de LILLE, Lille, Hauts-de-France, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Marino BS, Lipkin PH, Newburger JW, Peacock G, Gerdes M, Gaynor JW, Mussatto KA, Uzark K, Goldberg CS, Johnson WH Jr, Li J, Smith SE, Bellinger DC, Mahle WT; American Heart Association Congenital Heart Defects Committee, Council on Cardiovascular Disease in the Young, Council on Cardiovascular Nursing, and Stroke Council. Neurodevelopmental outcomes in children with congenital heart disease: evaluation and management: a scientific statement from the American Heart Association. Circulation. 2012 Aug 28;126(9):1143-72. doi: 10.1161/CIR.0b013e318265ee8a. Epub 2012 Jul 30. PMID 22851541
- [Result] Calderon J, Willaime M, Lelong N, Bonnet D, Houyel L, Ballon M, Goffinet F, Khoshnood B; EPICARD study group. Population-based study of cognitive outcomes in congenital heart defects. Arch Dis Child. 2018 Jan;103(1):49-56. doi: 10.1136/archdischild-2016-310830. Epub 2017 Aug 5. PMID 28780508
- [Result] Ryan KR, Jones MB, Allen KY, Marino BS, Casey F, Wernovsky G, Lisanti AJ. Neurodevelopmental Outcomes Among Children With Congenital Heart Disease: At-Risk Populations and Modifiable Risk Factors. World J Pediatr Congenit Heart Surg. 2019 Nov;10(6):750-758. doi: 10.1177/2150135119878702. Epub 2019 Oct 28. PMID 31658880
- [Result] Jayaram N, Spertus JA, Kennedy KF, Vincent R, Martin GR, Curtis JP, Nykanen D, Moore PM, Bergersen L. Modeling Major Adverse Outcomes of Pediatric and Adult Patients With Congenital Heart Disease Undergoing Cardiac Catheterization: Observations From the NCDR IMPACT Registry (National Cardiovascular Data Registry Improving Pediatric and Adult Congenital Treatment). Circulation. 2017 Nov 21;136(21):2009-2019. doi: 10.1161/CIRCULATIONAHA.117.027714. Epub 2017 Sep 7. PMID 28882885
- [Result] Mulkey SB, Yap VL, Bai S, Ramakrishnaiah RH, Glasier CM, Bornemeier RA, Schmitz ML, Bhutta AT. Amplitude-integrated EEG in newborns with critical congenital heart disease predicts preoperative brain magnetic resonance imaging findings. Pediatr Neurol. 2015 Jun;52(6):599-605. doi: 10.1016/j.pediatrneurol.2015.02.026. Epub 2015 Mar 5. PMID 25838043
- [Result] Mebius MJ, Kooi EMW, Bilardo CM, Bos AF. Brain Injury and Neurodevelopmental Outcome in Congenital Heart Disease: A Systematic Review. Pediatrics. 2017 Jul;140(1):e20164055. doi: 10.1542/peds.2016-4055. Epub 2017 Jun 13. PMID 28607205
- [Result] Asakai H, Cardamone M, Hutchinson D, Stojanovski B, Galati JC, Cheung MM, Mackay MT. Arterial ischemic stroke in children with cardiac disease. Neurology. 2015 Dec 8;85(23):2053-9. doi: 10.1212/WNL.0000000000002036. Epub 2015 Sep 25. PMID 26408496
- [Result] Latal B, Wohlrab G, Brotschi B, Beck I, Knirsch W, Bernet V. Postoperative Amplitude-Integrated Electroencephalography Predicts Four-Year Neurodevelopmental Outcome in Children with Complex Congenital Heart Disease. J Pediatr. 2016 Nov;178:55-60.e1. doi: 10.1016/j.jpeds.2016.06.050. Epub 2016 Jul 22. PMID 27453368
- [Result] Meyer S, Poryo M, Shatat M, Gortner L, Abdul-Khaliq H. The role of EEG recordings in children undergoing cardiac surgery for congenital heart disease. Wien Med Wochenschr. 2017 Sep;167(11-12):251-255. doi: 10.1007/s10354-017-0576-0. Epub 2017 Jun 28. PMID 28660303
- [Result] Shellhaas RA, Chang T, Tsuchida T, Scher MS, Riviello JJ, Abend NS, Nguyen S, Wusthoff CJ, Clancy RR. The American Clinical Neurophysiology Society's Guideline on Continuous Electroencephalography Monitoring in Neonates. J Clin Neurophysiol. 2011 Dec;28(6):611-7. doi: 10.1097/WNP.0b013e31823e96d7. No abstract available. PMID 22146359
- [Result] Gutierrez-Colina AM, Topjian AA, Dlugos DJ, Abend NS. Electroencephalogram monitoring in critically ill children: indications and strategies. Pediatr Neurol. 2012 Mar;46(3):158-61. doi: 10.1016/j.pediatrneurol.2011.12.009. PMID 22353290
- [Result] Peyvandi S, Chau V, Guo T, Xu D, Glass HC, Synnes A, Poskitt K, Barkovich AJ, Miller SP, McQuillen PS. Neonatal Brain Injury and Timing of Neurodevelopmental Assessment in Patients With Congenital Heart Disease. J Am Coll Cardiol. 2018 May 8;71(18):1986-1996. doi: 10.1016/j.jacc.2018.02.068. PMID 29724352
- [Result] Meuwly E, Feldmann M, Knirsch W, von Rhein M, Payette K, Dave H, Tuura ROG, Kottke R, Hagmann C, Latal B, Jakab A; Research Group Heart and Brain*. Postoperative brain volumes are associated with one-year neurodevelopmental outcome in children with severe congenital heart disease. Sci Rep. 2019 Jul 26;9(1):10885. doi: 10.1038/s41598-019-47328-9. PMID 31350426
- [Result] Claessens NHP, Khalili N, Isgum I, Ter Heide H, Steenhuis TJ, Turk E, Jansen NJG, de Vries LS, Breur JMPJ, de Heus R, Benders MJNL. Brain and CSF Volumes in Fetuses and Neonates with Antenatal Diagnosis of Critical Congenital Heart Disease: A Longitudinal MRI Study. AJNR Am J Neuroradiol. 2019 May;40(5):885-891. doi: 10.3174/ajnr.A6021. Epub 2019 Mar 28. PMID 30923087
- [Result] Long SH, Harris SR, Eldridge BJ, Galea MP. Gross motor development is delayed following early cardiac surgery. Cardiol Young. 2012 Oct;22(5):574-82. doi: 10.1017/S1047951112000121. Epub 2012 Feb 29. PMID 22373640
- [Result] Flamant C, Branger B, Nguyen The Tich S, de la Rochebrochard E, Savagner C, Berlie I, Roze JC. Parent-completed developmental screening in premature children: a valid tool for follow-up programs. PLoS One. 2011;6(5):e20004. doi: 10.1371/journal.pone.0020004. Epub 2011 May 26. PMID 21637833
- [Result] Ribera I, Ruiz A, Sanchez O, Eixarch E, Antolin E, Gomez-Montes E, Perez-Cruz M, Cruz-Lemini M, Sanz-Cortes M, Arevalo S, Ferrer Q, Vazquez E, Vega L, Dolader P, Montoliu A, Boix H, Simoes RV, Masoller N, Sanchez-de-Toledo J, Comas M, Bartha JM, Galindo A, Martinez JM, Gomez-Roig L, Crispi F, Gomez O, Carreras E, Cabero L, Gratacos E, Llurba E. Multicenter prospective clinical study to evaluate children short-term neurodevelopmental outcome in congenital heart disease (children NEURO-HEART): study protocol. BMC Pediatr. 2019 Sep 10;19(1):326. doi: 10.1186/s12887-019-1689-y. PMID 31506079
- [Result] Hirsch LJ, Fong MWK, Leitinger M, LaRoche SM, Beniczky S, Abend NS, Lee JW, Wusthoff CJ, Hahn CD, Westover MB, Gerard EE, Herman ST, Haider HA, Osman G, Rodriguez-Ruiz A, Maciel CB, Gilmore EJ, Fernandez A, Rosenthal ES, Claassen J, Husain AM, Yoo JY, So EL, Kaplan PW, Nuwer MR, van Putten M, Sutter R, Drislane FW, Trinka E, Gaspard N. American Clinical Neurophysiology Society's Standardized Critical Care EEG Terminology: 2021 Version. J Clin Neurophysiol. 2021 Jan 1;38(1):1-29. doi: 10.1097/WNP.0000000000000806. No abstract available. PMID 33475321
- [Result] Murray DM, Boylan GB, Ryan CA, Connolly S. Early EEG findings in hypoxic-ischemic encephalopathy predict outcomes at 2 years. Pediatrics. 2009 Sep;124(3):e459-67. doi: 10.1542/peds.2008-2190. Epub 2009 Aug 24. PMID 19706569
- [Result] Barkovich AJ, Hajnal BL, Vigneron D, Sola A, Partridge JC, Allen F, Ferriero DM. Prediction of neuromotor outcome in perinatal asphyxia: evaluation of MR scoring systems. AJNR Am J Neuroradiol. 1998 Jan;19(1):143-9. PMID 9432172
- [Result] Agarwal S, Sud K, Menon V. Nationwide Hospitalization Trends in Adult Congenital Heart Disease Across 2003-2012. J Am Heart Assoc. 2016 Jan 19;5(1):e002330. doi: 10.1161/JAHA.115.002330. PMID 26786543
- [Result] Lacour-Gayet F, Clarke D, Jacobs J, Gaynor W, Hamilton L, Jacobs M, Maruszewski B, Pozzi M, Spray T, Tchervenkov C, Mavroudis C; Aristotle Committee. The Aristotle score for congenital heart surgery. Semin Thorac Cardiovasc Surg Pediatr Card Surg Annu. 2004;7:185-91. doi: 10.1053/j.pcsu.2004.02.011. PMID 15283368
- [Result] Budts W, Borjesson M, Chessa M, van Buuren F, Trigo Trindade P, Corrado D, Heidbuchel H, Webb G, Holm J, Papadakis M. Physical activity in adolescents and adults with congenital heart defects: individualized exercise prescription. Eur Heart J. 2013 Dec;34(47):3669-74. doi: 10.1093/eurheartj/eht433. Epub 2013 Nov 7. No abstract available. PMID 24204010